CLINICAL TRIAL: NCT04152954
Title: Comparison of a Multi-tined Cannula Versus a Conventional Cannula for Cervical Medial Branch Radiofrequency Ablation in Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19.101
Record Dates: First submitted 2019-11-01; First posted 2019-11-06 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Neck Pain; Radiofrequency Ablation; Facet Joint Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional cannula (Active Comparator): Cervical Medial Branch Radiofrequency Neurotomy using a conventional cannula, the patient lying prone with a posterior approach.
  Interventions: Device: Radiofrequency ablation of cervical medial branches
- Multi-tined cannula (Experimental): Cervical Medial Branch Radiofrequency Neurotomy using a Multi-Tined cannula, the patient lying in lateral decubitus with a lateral approach
  Interventions: Device: Radiofrequency ablation of cervical medial branches

INTERVENTIONS:
Device: Radiofrequency ablation of cervical medial branches — Radiofrequency ablation of cervical medial branches

SUMMARY:
Chronic neck pain is a common disorder for spine specialists. Radiofrequency ablation of medial branches has been proven effective in selected patients for relieving pain. A newer radiofrequency ablation cannula has been developed (multi-tined), allowing perpendicular access. It is proposed as an alternative to the more technically challenging traditional approach. This study aims to compared the technical and clinical aspects of both techniques.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Cervical neck pain at least 4/10 at rest or with activity
* Neck pain lasting at least 6 months and refractory to conservative treatments
* Neck pain is primarily axial (more than upper extremity)
* Success to medial branch block protocol

Exclusion Criteria:

* failure to medial branch block protocol (pain relief less than 75% on 2 occasions)
* Cervical neck pain less than 4/10
* Neurological deficits of upper extremity
* neuropathic pain of upper extremity
* pregnancy or breastfeeding
* inflammatory or neoplastic lesion on x-ray
* neck cortisone injection in last 3 months
* any medical or psychiatric condition contra-indicated for radiofrequency ablation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Rating scale for patient's pain during the procedure | 1 day of the intervention
  pain during radiofrequency procedure will be compared between the 2 groups as a principal hypothesis is that the new multi-tined cannula is better tolerated by patients Scale is from 0-10, 0/10 is no pain which is better than pain of 10/10

SECONDARY OUTCOMES:
Fluoroscopy time | 1 day of the intervention
  Calculated time of fluoroscopy in seconds
Radiation dosage | 1 day of the intervention
  Calculated dose of radiation measure by the C-arm
time of procedure | 1 day of the intervention
  Total time of procedure in minutes/seconds
Patient pain (Numerical Rating Scale - NRS score) | 0, 3, 6 12 months
  therapeutic effect on pain Scale is from 0-10, 0/10 is no pain which is better than pain of 10/10
Patient function (Neck disability Index - NDI) | 0, 3, 6, 12 months
  therapeutic effect on function scale is from 0-100%, where 0% is better than 100% in terms of the effect of pain on function

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No